CLINICAL TRIAL: NCT07257497
Title: Safety and Efficacy of Combining a Vitamin B6-Limited Diet With Immunotherapy in Solid Tumor Patients: A Clinical Study Protocol
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xuelei Ma MD, Department of Biotherapy, Cancer Center and State Key Laboratory of Biotherapy, West China Hospital, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Approval No. 1069 (2025)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor Cancer
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Intervention Model Description: Vitamin B6-restricted Diet
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Vitamin B6-restricted diet + immunotherapy (Experimental)
  Interventions: Dietary Supplement: Vitamin B6-restricted diet + immunotherapy

INTERVENTIONS:
Dietary Supplement: Vitamin B6-restricted diet + immunotherapy — Targeted Vitamin B6 Metabolism: The intervention zeroes in on Vitamin B6 metabolism. As solid tumors often have Vitamin B6 synthesis flaws and rely on external Vitamin B6, dietary restriction of Vitamin B6 is a novel approach. Dietary Intervention: The -vitB6 liquid diet in this study is precisely defined. Dosage is determined by patient weight, following 30 kcal/kg/day for energy and 1.5 g/kg/day for protein. A low -vitB6 food list is provided. Study Design and Endpoints: It's a Phase I single - arm study. Its main goal is to evaluate the safety and tolerance of the combined treatment. Secondary and exploratory endpoints cover efficacy, nutritional state, and immune status.

SUMMARY:
This is a phase I single-arm clinical study conducted by West China Hospital of Sichuan University. The research duration is from October 2025 to June 2027, aiming to evaluate the safety and efficacy of vitamin B6-restricted (-VitB6 diet) in patients with solid tumors. A total of 20 patients with solid tumors, aged 18 - 75 years old, who meet specific inclusion criteria such as having at least one measurable lesion according to RECIST v1.1 criteria and an ECOG score of 0 - 1, will be enrolled.

Patients will receive -VitB6 diet intervention for 2 cycles (3 weeks per cycle) while continuing their original immunotherapy. The -VitB6 diet strictly limits vitamin B6 intake, and patients can only consume foods with extremely low vitamin B6 content. The research will collect data on patients' basic information, nutritional status, blood, immunity, and tumor imaging at baseline and during follow - up.

The primary endpoint of the study is the occurrence type, frequency, and severity of treatment-related adverse events (TEAE). Secondary endpoints include objective response rate (ORR), disease control rate (DCR), and duration of response (DoR). Exploratory endpoints involve evaluating the nutritional adequacy of the -VitB6 diet, its impact on patients' quality of life, and its influence on amino acid metabolism and immune status in patients.

During the study, safety will be evaluated by closely monitoring adverse events according to NCI CTCAE (version 5.0), and efficacy will be assessed using RECIST 1.1 standard. Statistical analysis will be performed using SAS 9.4 software, including descriptive statistics for safety and efficacy data, and calculating confidence intervals for relevant indicators. This study hopes to provide new strategies and directions for the treatment of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* (1) Sign a written informed consent form before any study - related procedures are carried out.

  (2) Males or females, aged 18 - 80 years old. (3) Diagnosed with solid tumors by pathological tissue biopsy. (4) According to the RECIST v1.1 (Response Evaluation Criteria in Solid Tumors Version 1.1) criteria, there is at least 1 measurable lesion (lesions previously treated with local therapies such as radiotherapy cannot be regarded as measurable lesions).

  (5) ECOG (Eastern Cooperative Oncology Group Performance Status) score of 0 - 1.

  (6) NRS - 2002 (Nutritional Risk Screening 2002) score < 3. (7) BMI (Body Mass Index) ≥ 18.5 (can be adjusted appropriately according to the actual situation).

  (8) Patients who can eat orally or through a feeding tube and can tolerate enteral nutrition.

  (9) Sufficient organ function, and the subjects need to meet the following laboratory indicators: In the absence of granulocyte - colony - stimulating factor use in the past 14 days, the absolute neutrophil count ≥ 1.5×10⁹/L.

Platelets ≥ 75×10⁹/L. In the absence of blood transfusion or erythropoietin use in the past 7 days, hemoglobin ≥ 8 g/dL.

Serum albumin ≥ 3.0 g/dL. Total bilirubin ≤ 1.5× the upper limit of normal (ULN). Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5×ULN. In case of liver metastasis, ALT and/or AST ≤ 5×ULN, and total bilirubin ≤ 3×ULN. In case of liver or bone metastasis, Alkaline Phosphatase (AKP) ≤ 5×ULN.

Creatinine clearance rate ≥ 50 mL/min (calculated according to the Cockcroft - Gault formula) or serum creatinine ≤ 1.5×ULN.

International Normalized Ratio (INR) ≤ 1.5×ULN, Prothrombin Time (PT) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5×ULN.

Urine protein < 2+ (if urine protein ≥ 2+, a 24 - hour urine protein quantification can be performed, and subjects with a 24 - hour urine protein quantification < 2.0 g can be enrolled).

(10) Women of child - bearing potential must agree to avoid sexual intercourse (heterosexual intercourse) or use a reliable and effective contraceptive method from the signing of the informed consent form until at least 6 months after the last administration of the study drug. In addition, the serum HCG (Human Chorionic Gonadotropin) test must be negative within 3 days before the start of the study treatment, and the subject must be non - lactating. A female patient is considered to be of child - bearing potential if she is post - menopausal but has not reached the post - menopausal state (non - menstrual period ≥ 12 consecutive months, and no other causes are found except menopause) and has not undergone sterilization surgery (such as hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).

(11) If there is a risk of pregnancy, all subjects (regardless of male or female) need to use a contraceptive method with an annual failure rate of less than 1% throughout the treatment period until 120 days after the last administration of the study drug (or 180 days after the last administration of the chemotherapy drug).

Exclusion Criteria:

* (1) Patients with cognitive impairment or mental illness who are unable to understand the study content.

  (2) Patients with central nervous system or meningeal metastases. (3) Patients with clinically symptomatic moderate or severe ascites (that is, those who require therapeutic paracentesis within 2 weeks before the start of study treatment; patients with only a small amount of ascites shown on imaging and no clinical symptoms can be enrolled).

  (4) Patients with uncontrolled or moderate to severe pleural effusion and pericardial effusion.

  (5) Patients with severe diarrhea, intractable vomiting, severe malabsorption syndrome, paralytic and mechanical intestinal obstruction; tracheoesophageal fistula, gastrointestinal perforation or gastrointestinal fistula, or abdominal abscess; patients with extra - gastrointestinal bleeding with a CTCAE (Common Terminology Criteria for Adverse Events) grade 3 or above within 6 months before the start of study treatment or grade 2 or above within 3 months (such as abnormal vaginal bleeding, hematemesis).

  (6) Patients known to be allergic to the active ingredients or excipients of the study drug.

  (7) Patients with poorly controlled diabetes. (8) Patients with poorly controlled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg under routine antihypertensive treatment), with a history of hypertensive crisis or hypertensive encephalopathy.

  (9) Patients with severe cardiovascular and cerebrovascular diseases, including cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction, and major vascular diseases within 6 months before enrollment (including but not limited to aortic aneurysms requiring surgical repair or recent arterial thrombosis); patients with poorly controlled clinical symptoms or heart diseases, such as unstable angina pectoris, NYHA (New York Heart Association) heart failure grade II or above, left ventricular ejection fraction < 50% on color Doppler echocardiography, or severe arrhythmias that cannot be controlled by drug treatment.

  (10) Pregnant or lactating women. (11) Other situations considered by the investigator as inappropriate for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-09 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of Vitamin B6 restricted diet (-Vit B6 diet) combined with immunotherapy in patients with solid tumors. | From enrollment to the end of treatment at 6 weeks
  The occurrence types, frequencies, and severities of treatment - emergent adverse events (TEAE).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From enrollment to the end of treatment at 1 year
  Evaluate the effectiveness of Vitamin B6-restricted diet combined with immunotherapy in patients with solid tumors.
Disease Control Rate (DCR) | From enrollment to the end of treatment at 1 year
  Evaluate the effectiveness of Vitamin B6-restricted diet combined with immunotherapy in patients with solid tumors.
Duration of Response (DoR) | From enrollment to the end of treatment at 1 year
  Evaluate the effectiveness of Vitamin B6-restricted diet combined with immunotherapy in patients with solid tumors.

IPD SHARING:
Plan to Share IPD: No